CLINICAL TRIAL: NCT06889636
Title: Assessment of the Impact of Pharmaceutical Care on the Quality of Life in Conditions Related to Psychotropic Drug Use and Evaluation of the Intervention
Brief Title: Pharmaceutical Care and Quality of Life in Conditions Related to Psychotropic Drug Use
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rijeka (Other)
Responsible Party: Principal Investigator, Alena Tatarevic, Assessment of the impact of pharmaceutical care on the quality of life in conditions related to psychotropic drug use and evaluation of the intervention, University of Rijeka
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 200-07/2023-01/1_001/2023
Record Dates: First submitted 2025-02-25; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-02

CONDITIONS: Mental Health Services
Keywords: Mental disorders; Quality of life; Drug-related problems
MeSH Terms: conditions — Mental Disorders | interventions — Pharmaceutical Services

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standardized pharmaceutical care (Experimental): Participants in group A received pharmacists' interventions based on standardized Medication Review (MR) and Medication Therapy Management (MTM) protocols.
  Interventions: Other: Pharmaceutical care in solving drug-related problems in subjects using psychotropic medicines based on standardized protocol..
- Basic counseling (Active Comparator): Participants enrolled in group B received pharmaceutical care based on common pharmacist´s practice in Croatia.
  Interventions: Other: Common pharmacists' practice in Croatia.

INTERVENTIONS:
Other: Pharmaceutical care in solving drug-related problems in subjects using psychotropic medicines based on standardized protocol.. — Pharmacists' interventions were based on Medication Review and Medication Therapy Management evaluations of a subjects' pharmacotherapy to optimize medicine use, improve treatment outcomes and quality of life. The intervention involved the identification of drug-related problems and addressing these issues through pharmacist interventions. The intervention was based on information gathered from the subjects and a list of medicines in use.
  Arms: Standardized pharmaceutical care
Other: Common pharmacists' practice in Croatia. — Group B participants received pharmaceutical care based on common pharmacists' practice in Croatia during the dispensing of psychotropic drugs.
  Arms: Basic counseling

SUMMARY:
This study aims to assess and describe the impact of pharmaceutical care on identified drug-related problems (DRPs) in subjects using psycholeptics and psychoanaleptics in primary care, improving subjects' self-assessed quality of life (QoL)

The hypothesis of the study are:

1. Side-effects are the most common DRPs in subjects using psychotropic medicines in primary care,
2. Treatment effectiveness and safety affect the subjects´ QoL

DETAILED DESCRIPTION:
The study objectives are to:

1. assess QoL in subjects using psycholeptics and psychoanaleptics,
2. analyze identified DRPs and their causes in subjects using psycholeptics and psychoanaleptics
3. evaluate the correlation between the type and total number of DRPs identified in a single subject with QoL,
4. describe the impact of pharmacists´ intervention in the identification and resolution of the DRPs and their causes on subjects´ QoL.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants (years 18+)
* Usage of psycholeptic or psychoanaleptic medicines
* Residence in Istrian County (Croatia)

Exclusion Criteria:

* Minor participants
* Hospitalization during study participation
* Unable to live by themselves
* Unable to participate in study for 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2025-02-14 (Actual); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Assessment of the quality of life in subjects using psycholeptics and psychoanaleptics | Prior and after the pharmacists' intervention during three months period.
  A short version of the World Health Organization's quality of life questionnaire (WHOQOL-BREF questionnaire) is being used to assess subjects' QoL. The scale range is from 0 to 100. A higher score number indicates better QoL.

SECONDARY OUTCOMES:
Analysis of identified drug-related problems | During period of three months.
  To analyze the type of DRPs, validated Classification for Drug-Related Problems from the Pharmaceutical Care Network Europe Association, version 9.1 has been used. PCNE Classification for DRPs describes each type of DRP by unique code.

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmacy Bobanovic Vujnovic Pula, Pula, Croatia

IPD SHARING:
Plan to Share IPD: No